CLINICAL TRIAL: NCT00810134
Title: A Randomised Controlled Trial for the Treatment of 5 - 25 cm Superficial Femoral Artery oc-Clusions Comparing Femoropopliteal Bypass With 6 mm PTFE-Prosthesis and 6 - 7 mm Viabahn Endoprosthesis
Brief Title: Bypass or Thurpass for Superficial Femoral Artery Occlusion? Scandinavian Thurpass Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the results of interim analysis at the time 44 patients were recruited.
Sponsor: University of Helsinki (Other)
Collaborators: W.L.Gore & Associates (Industry)
Responsible Party: Mauri Lepantalo, Department of Vascular Surgery, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Version 1.7 - Oct 15th 2002
Record Dates: First submitted 2008-12-15; First posted 2008-12-17 (Estimated); Last update posted 2008-12-17 (Estimated); Status verified 2008-12

CONDITIONS: Femoral Artery Occlusion
Keywords: Superficial femoral artery occlusion (TASC II B or C)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thrupass (Other): Endovascular treatment (Thrupass) is performed as a femoropopliteal above knee endovascular recanalisation and Viabahn introduction with 6-7 mm Viabahn endo-prosthesis.
  Interventions: Procedure: Thrupass
- Bypass (Other): Surgical procedure is performed as a femoropopliteal above knee by-pass with 6 mm non-coated PTFE-graft
  Interventions: Procedure: Bypass

INTERVENTIONS:
Procedure: Thrupass — Endovascular treatment (Thrupass) is performed as a femoropopliteal above knee endovascular recanalisation and Viabahn introduction with 6-7 mm Viabahn endo-prosthesis.
  Arms: Thrupass
Procedure: Bypass — Surgical procedure is performed as a femoropopliteal above knee by-pass with 6 mm non-coated PTFE-graft
  Arms: Bypass

SUMMARY:
The aim of the study is to compare PTFE-graft bypass surgery versus Viabahn endoprosthesis for femoropopliteal arterial occlusion in intermittent claudication and critical ischaemia in patients who would be technically amenable for both treatments. The primary objective is to compare primary patencies of the two treatments. The secondary objective of the study is to evaluate secondary patency, functional status, the quality of life and costs of the new endovascular therapy.

DETAILED DESCRIPTION:
Femoropopliteal bypass graft surgery with PTFE-prosthesis has proven to be an acceptable treatment for stable incapacitating claudication and critical ischaemia in patients with superficial femoral artery occlusion. Preliminary results of a thrupass endoprosthesis in the treatment of femoral lesions are promising. Less morbidity and better cost-effectiveness are suggested to be achieved in treatment of chronic lower limb ischaemia with endovascular treatment comparing to surgical treatment.

A randomised multicentre trial aims to enrol a pilot group of 60 + 60 patients to be followed for 3 years. Patients are treated either with Viabahn thrupass endoprosthesis (Gore corp.) or with 6 mm PTFE-prosthesis bypass graft surgery. Primary patency at three years is the primary end point and secondary patency, functional success, costs and quality of life are the secondary end points.

ELIGIBILITY:
Inclusion Criteria:

1. Superficial femoral artery occlusion from 5 to 25 cm in length above the knee joint.
2. Patient must be equally eligible for both procedures.
3. Patient must present intermittent claudication with resistance to medical therapy and exercise or critical ischaemia.
4. Normal adjacent vessel diameter must be between 4.8 and 6.5 mm.
5. At least one patent distal run-off vessel and at least 1 cm of healthy superficial femoral artery below and above the lesion to allow proper placement of the endoprosthesis.
6. Patient must be 18 years or older.
7. Women of childbearing age must have negative pregnancy test prior to inclusion.

Exclusion Criteria:

1. Known allergy or contraindications to aspirin, clopidogrel, dipyridamole or anticoagulants.
2. Bleeding diatheses
3. Presence of one or several previously placed endoprosthesis or grafts in the superficial femoral artery segment.
4. Planned other endovascular therapy of the same segment.
5. Other than 6-7 mm diameter endoprosthesis or 6 mm PTFE-prosthesis is needed.
6. Presence of evolving malignant cancer or any other illness posing an immediate threat to life.
7. Life-expectancy less than 2 years due to co-morbidity or other situation that would make the patient unlikely candidate for follow-up visits.
8. Participation in another vascular clinical study less than 30 days prior to inclusion.
9. Patients unable to fill out the prescribed quality of life questionnaires themselves or unable to understand the full meaning of the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2003-01; Primary Completion 2008-02 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Primary end point of the study will be primary patency. Patency should be demonstrated by duplex ultrasound or other imaging modality at every control visit. ABI measurements will be recorded to assess the haemodynamic effect of the procedure. | At three years after intervention

SECONDARY OUTCOMES:
Suboptimal outcome is defined as the presence of any of the following: re-stenosis diagnosed by colour duplex ultrasonography, ankle-brachial index improvement of less than 0.15, or re-intervention at the treated site. | At any time of the study
Secondary patency is defined by procedures required to re-establish or maintain blood flow after occlusion. | At any time of the study
Complications will include post procedure haemorrhage, haematomas, cardiac, pulmonary and renal complications and infection. Technical problems or equipment failure in the endoprosthesis group will also be recorded. | At any time of the study
A procedural death will be any death that will occur within 30 days of the procedure. | At any time of the study
Immediate functional failure is one in which the threshold increase of ABI is not achieved within 24 hours. Early failure is any failure occurring within 30 days of the operation. | within 30 days of the operation
Limb salvage is defined as retention of the leg without any major amputation or death. | At any time of the study

CONTACTS AND LOCATIONS:
Overall Officials: Mauri Lepantalo, M.D., PhD, Principal Investigator — Department of Vascular Surgery, Helsinki University Central Hospital
Locations (1):
- Department of Vascular Surgery, Helsinki University Central Hospital, Helsinki, Finland